CLINICAL TRIAL: NCT03289234
Title: A Multi-Center, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics of MCI-186 in Subjects With Mild or Moderate Hepatic Impairment Compared to Subjects With Normal Hepatic Function
Brief Title: Pharmacokinetics Study of MCI-186 in Subjects With Mild or Moderate Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MCI-186-J23
Record Dates: First submitted 2017-09-19; First posted 2017-09-20 (Actual); Results first posted 2020-02-28 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Hepatic Impairment; Healthy
MeSH Terms: interventions — Edaravone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mild hepatic impairment (Experimental)
  Interventions: Drug: MCI-186
- moderate hepatic impairment (Experimental)
  Interventions: Drug: MCI-186
- normal hepatic function (Experimental)
  Interventions: Drug: MCI-186

INTERVENTIONS:
Drug: MCI-186 — 30 mg of edaravone will be administered intravenously over 60 minutes
  Other Names: Edaravone; Radicut

SUMMARY:
To assess the pharmacokinetics of MCI-186 after a single intravenous infusion of 30mg/hour in subjects with mild or moderate Hepatic impairment compared to subjects with normal hepatic function

ELIGIBILITY:
Inclusion Criteria:

All subjects

* Able to provide written informed consent to participate in this study after reading the ICF
* Subjects is able to understand and willing to cooperate and comply with the Protocol restrictions and requirements.
* A body weight of ≥45 kg in males or ≥40 kg in females and a body mass index ranging from 18 to 30 kg/m2

Hepatic impaired subjects (in addition)

* A Child-Pugh score of 5 or 6 for subjects with mild hepatic impairment, and between 7 and 9, inclusive, for subjects with moderate hepatic impairment
* Chronic and stable hepatic impairment

Healthy subjects (in addition)

* Subject with normal hepatic function
* Good health and free from clinically significant illness or disease

Exclusion Criteria:

All subjects

* Presence or history of severe allergy to food, or any medicinal product or relevant excipient that is of clinical significance
* Subjects were previously administered MCI-186.
* Positive urine drug screen (if not due to concomitant medication) or alcohol test
* History of drug abuse
* Presence of alcohol abuse
* Presence of active infection requiring antibiotics
* Positive test for human immunodeficiency virus (HIV) antigen/antibody
* Uncontrolled, or untreated hypertension defined as systolic blood pressure (SBP)>160 mmHg and/or diastolic blood pressure (DBP)>100 mmHg
* eGFR <60 mL/min/1.73m2

Hepatic impairment subject (in addition)

* Subjects with severe ascites

Healthy subject (in addition)

* History or presence of any parenchymal hepatic disease
* Positive test for hepatitis B surface antigen (HBsAg) and hepatitis C virus antibody (HCVAb)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (2):
- Japan (2):
  - Investigational site, Fukuoka
  - Investigational site, Tokyo

REFERENCES:
- [Derived] Nakamaru Y, Kakubari M, Yoshida K, Akimoto M, Todorovic V, Greis T, Kondo K. Open-label, Single-dose Studies of the Pharmacokinetics of Edaravone in Subjects with Mild, Moderate, or Severe Hepatic Impairment Compared to Subjects with Normal Hepatic Functioning. Clin Ther. 2020 Aug;42(8):1467-1482.e4. doi: 10.1016/j.clinthera.2020.06.016. Epub 2020 Aug 14. PMID 32800532

RESULTS

PARTICIPANT FLOW:
Groups:
- Mild Hepatic Impairment: Child-Pugh score of 5 or 6
- Moderate Hepatic Impairment: Child-Pugh score between 7 and 9
- Normal Hepatic Function: normal hepatic function
Period: Overall Study
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Normal Hepatic Function
Started | 8 | 6 | 8
Completed | 8 | 6 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Normal Hepatic Function | Total
Number analyzed (Participants) | 8 | 6 | 8 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (11.9) | 66.2 (5.3) | 61.6 (2.7) | 62.1 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 5
  Male | 6 | 5 | 6 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 8 | 6 | 8 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Time Frame: pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 6 | 8
ng/mL | 538.1 (182.3) | 533.4 (88.57) | 429 (44.36)

2. Primary Outcome: AUC0-last
Time Frame: pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 6 | 8
ng*hr/mL | 716.86 (258.3) | 739.28 (146.89) | 582.89 (58.33)

3. Primary Outcome: AUC0-∞
Time Frame: pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 6 | 8
ng*hr/mL | 727.55 (262.04) | 751.52 (148.34) | 594.96 (63.58)

4. Secondary Outcome: t½
Time Frame: pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 6 | 8
hour | 3.14 (0.58) | 4.37 (1.9) | 5.41 (6.58)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Normal Hepatic Function
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 1/6 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mild Hepatic Impairment (N=8) | Moderate Hepatic Impairment (N=6) | Normal Hepatic Function (N=8)
Chest pain (General disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT03289234/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT03289234/SAP_001.pdf